CLINICAL TRIAL: NCT06162377
Title: Methylnatrexone In Resectable Head and Neck Squamous Cell Carcinoma (MINK). A "Window of Opportunity" Pilot Study.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0729; NCI-2023-10299 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — methylnaltrexone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Methylnaltrexone (Experimental): Participants will be given 14 pre-filled syringes of methylnaltrexone. Participants will be instructed how to take the drug as an injection under the skin of your abdominal area.
  Interventions: Drug: Methylnaltrexone

INTERVENTIONS:
Drug: Methylnaltrexone — Given by SC (injection)
  Other Names: Relistor™

SUMMARY:
To learn if OCSCC patients can be safely given methylnaltrexone for 2 weeks before surgery.

DETAILED DESCRIPTION:
2.1 Primary Objectives

The primary objective of this study is to evaluate the feasibility of treating OCSCC participants with methylnaltrexone. We define success as when a participants can receive assigned medication for two weeks preoperatively without interruption due to AEs (NCI CTCAE v4.03). By the end of the trial, feasibility is claimed if 90% or above the participants can successfully receive assigned medication.

2.2 Secondary Objectives

The secondary objectives are to evaluate the endpoints include tolerability, efficacy and tumor biological response of methylnaltrexone in surgical candidates for OCSCC.

2.3 Exploratory Objectives

The exploratory objectives are to perform tumor RNASeq profiling and assess blood and tumor immunological landscape, and to correlate efficacy endpoints with tumor biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older. Because no dosing or adverse event data are currently available on the use of methylnaltrexone in participants <18 years of age, children are excluded from this study.
* Histologically-confirmed oral cavity squamous cell carcinoma [(T1-T4, N (any)] that is amenable to curative-intent surgery
* Able to receive the study drug for at least two weeks preoperatively
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures
* The effects of methylnaltrexone on the developing human fetus are unknown. For this reason and because methylnaltrexone agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. This includes all female participants, between the onset of menses (as early as 8 years of age) and 55 years unless the participants presents with an applicable exclusionary factor which may be one of the following:

  * Postmenopausal (no menses in greater than or equal to 12 consecutive months).
  * History of hysterectomy or bilateral salpingo-oophorectomy.
  * Ovarian failure (Follicle Stimulating Hormone and Estradiol in menopausal range, who have received Whole Pelvic Radiation Therapy).
  * History of bilateral tubal ligation or another surgical sterilization procedure.
  * Approved methods of birth control are as follows: Hormonal contraception (i.e. birth control pills, injection, implant, transdermal patch, vaginal ring), Intrauterine device (IUD), Tubal Ligation or hysterectomy, Subject/Partner post vasectomy, Implantable or injectable contraceptives, and condoms plus spermicide. Not engaging in sexual activity for the total duration of the trial and the drug washout period is an acceptable practice; however periodic abstinence, the rhythm method, and the withdrawal method are not acceptable methods of birth control. Should a woman become pregnant or suspect she is pregnant while her partner participates in this study, she should inform her treating physician immediately.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* Non-English/Non-Spanish speaking participants.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to methylnaltrexone or other agents used in the study.
* Participants with uncontrolled intercurrent illness, including chronic kidney disease defined as a eGRF <60 ml/mim, and liver disease defined as transaminitis > 2 folds from normal levels, cirrhosis and hyperbilirubinemia > 2 folds from normal levels
* Human immunodeficiency virus (HIV)-infected participants on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial.
* Participants with psychiatric illness/social situations that would limit compliance with study requirements.
* Urgent or emergency surgery
* Participants with known distant metastatic disease
* Participants with primary brain tumors or brain metastases. Methylnaltrexone has poor penetration of the blood brain barrier and there is limited available data regarding the safety of the drug in participants with central nervous system tumors.
* Pregnant women are excluded from this study because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with methylnaltrexone, breastfeeding should be discontinued if the mother is treated with methylnaltrexone. These potential risks may also apply to other agents used in this study.
* Peptic ulcer or intestinal perforation or colitis or other intestinal disorders such as Crohn's disease, diverticulitis, or Ogilvie's syndrome, intestinal obstruction or severe diarrhea because of risk of intestinal perforation.
* Use of other opioid antagonists because of the potential for additive effects of opioid receptor antagonism and increased risk of opioid withdrawal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and adverse events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Juan Cata, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org